CLINICAL TRIAL: NCT06117878
Title: An Open, Single Center Exploratory Study to Evaluate Safety and Efficacy of NK510 for Patients With Osteosarcoma and Soft Tissue Sarcoma
Brief Title: Safety and Efficacy of NK510 to Treat Osteosarcoma and Soft Tissue Sarcoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Base Therapeutics (Shanghai) Co., Ltd. (Industry)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NK510-05
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Osteosarcoma; Soft Tissue Sarcoma
MeSH Terms: conditions — Osteosarcoma; Sarcoma

STUDY DESIGN:
Intervention Model Description: Dose escalation study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A(low-dose group) (Experimental): NK510 1×10^9 NK cells/dose.
  Interventions: Drug: NK510
- Group B(medium-dose group) (Experimental): NK510 3×10^9 NK cells/dose.
  Interventions: Drug: NK510
- Group C(high-dose group) (Experimental): NK510 9×10^9 NK cells/dose.
  Interventions: Drug: NK510
- Group D(high-dose group，postoperative adjuvant treatmen) (Experimental): NK510 9×10^9 NK cells/dose.
  Interventions: Drug: NK510

INTERVENTIONS:
Drug: NK510 — NK510 will be administered through intravenous infusion.once a week，for a total of six times.
  Arms: Group A(low-dose group)
Drug: NK510 — NK510 will be administered through intravenous infusion.Twice infusions on week 1,week 3,week 5 respectively.
  Arms: Group B(medium-dose group); Group C(high-dose group); Group D(high-dose group，postoperative adjuvant treatmen)

SUMMARY:
This study will evaluate the safety and efficacy of NK510 in the treatment of Osteosarcoma and Soft Tissue Sarcoma.NK510 will be administered by intravenous injection. The safety and efficacy of this treatment will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent obtained,can be followed upon protocol;
* age ≥ 10 years;
* histopathologically confirmed diagnosis of advanced metastatic osteosarcoma or non-specific soft tissue sarcoma;
* Subjects for dose-escalation studies: failed to at least one chemotherapy regimen and undergoing disease progression or untolerable drug toxicity before enrollment;Subjects for postoperative adjuvant therapy study: radical surgery within 3 months before the first infusion of NK510 and no local recurrence or distant metastasis;
* according to RECIST 1.1,Recurrent and refractory patients have at least one measurable lesion at baseline. Patients receiving adjuvant treatment after radical surgery have no measurable lesions on imaging examination;
* ECOG physical status score of 0 or 1;
* Expected survival >=12 weeks;
* Female subjects of childbearing age or male subjects whose sexual partners are female subjects of childbearing age are required to take effective contraceptive measures throughout the entire treatment period and 6 months after the treatment period;
* good organ and bone marrow hematopoietic function, the laboratory test values within 7 days before enrollment meet the following requirements (no medication for blood components, cell growth factors, or albumin correction treatment is allowed within the first 14 days of obtaining laboratory test), as follows:

  1. Hematological:Neutrophil count ≥1.5×10^9/L; Platelet count ≥ 75×10^9/L; Hemoglobin ≥ 9 g/dL;
  2. Hepatic:Total bilirubin ≤1.5 x ULN;ALT and AST≤2.5×ULN;Albumin ≥ 28 g/L; Alkaline phosphatase ≤ 5 × ULN;
  3. Renal:Serum creatinine ≤ 1.25 × ULN or creatinine clearance ≥ 50mL/min (Cockcroft Fault formula);Patients whose urine routine results show urinary protein<2+or whose baseline urine routine test shows urinary protein ≥ 2+will undergo 24-hour urine collection with a 24-hour urine protein quantification of<1g.
  4. Coagulation:International standardized ratio (INR) ≤ 2, and activated partial thromboplastin time ≤ 1.5 × ULN.

Exclusion Criteria:

* Have received local or systemic anti-tumor treatment within 4 weeks before the first administration of NK510(Chinese medicine or traditional Chinese patent medicines and simple preparations is 2 weeks before administration);
* Untreated active hepatitis B (HbsAg positive and peripheral blood HBV-DNA>1000 IU/ml); Hepatitis C virus antibody positive;
* Patients with central nervous system metastasis;
* Previous history of arterial and venous thromboembolism events, including myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis, or any other serious thromboembolism within 6 month before NK510 first infusion;
* Severe bleeding tendency or coagulation dysfunction, or undergoing thrombolytic therapy;
* Uncontrolled hypertension, with systolic blood pressure ≥ 150mmHg or diastolic blood pressure ≥ 100mmHg after optimal medical treatment, hypertension crisis or history of hypertensive encephalopathy;
* Symptomatic congestive heart failure (New York Heart Association classification II-IV). Symptomatic or poorly controlled arrhythmia. The QT interval is prolonged, with QTc>450ms for males and 470ms for females. The echocardiography shows that the left ventricular ejection fraction at rest is less than 50%;
* Active pulmonary tuberculosis (TB), who is receiving anti-tuberculosis treatment or has received anti-tuberculosis treatment within one year before the first study medication;
* People infected with human immunodeficiency virus (HIV), known as active syphilis carriers;
* Severe infections that are active or poorly controlled clinically. Severe infection within 4 weeks prior to initial administration, including but not limited to hospitalization due to complications such as infection, bacteremia, or severe pneumonia;
* Administer therapeutic antibiotics orally or intravenously within one week before starting the study treatment;
* Active autoimmune diseases requiring systemic treatment have occurred within 2 years prior to the first administration. Allow the use of alternative therapies (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency). A known history of primary immunodeficiency;
* Within 4 weeks before the first administration, immunosuppressive drugs have been used, excluding local corticosteroids administered through nasal spray, inhalation, or other means, or systemic corticosteroids administered in physiological doses (i.e. no more than 10 mg/day of prednisone equivalent dose). Temporary use of corticosteroids is allowed for the prevention of allergic reactions or the treatment of respiratory distress symptoms such as asthma and chronic obstructive pulmonary disease;
* Within 4 weeks before the first administration or planned to receive live attenuated vaccines during the study period;
* Uncontrolled/uncorrectable metabolic disorders or other non malignant tumor organ diseases or systemic diseases or secondary reactions to cancer, which can lead to high medical risk and/or uncertainty in survival evaluation;
* Other acute or chronic diseases, mental illnesses, or abnormal laboratory test values that may lead to increased risk of study participation or drug administration, or interference with the interpretation of study results, based on the judgment of the investigator, the patient is not eligible to participate in this study;
* Diagnosed as other malignant tumors within 5 years prior to the first administration, excluding basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or carcinoma in situ after radical resection;
* Those who have participated in clinical trials of other drugs and received treatment with investigational drugs within 4 weeks before the first administration;
* Within 2 weeks before the first administration, medication with immunomodulatory effects (including thymosin, interferon, interleukin, except for local use to control pleural or ascites) has been received;
* Pregnant or lactating female patients.

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity | 6 weeks
  To evaluate the DLT during N510 treatment
Maximal Tolerable Dose | 6 weeks
  To evaluate the MTD of NK510

SECONDARY OUTCOMES:
Overall response rate (ORR) | 6 weeks
  Effectiveness Metrics

CONTACTS AND LOCATIONS:
Overall Officials: Yingqi Hua, phD, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No